CLINICAL TRIAL: NCT04069780
Title: Comparative Study Between Intravitreal and Suprachoroidal Injection of Triamcinolone Acetonide for Management of Diabetic Macular Edema
Brief Title: Suprachoroidal Injection of Triamcinolone Acetonide for Management of Diabetic Macular Edema
Acronym: SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azza Mohamed Ahmed Said (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Azza Mohamed Ahmed Said, Professor of Ophthalmology, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AinShamsU1
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Safety; Efficacy
Keywords: Suprachoroidal injection; Diabetic macular edema; Tiamicinolone acetonide
MeSH Terms: interventions — Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group I : Intravitreal injection (Active Comparator): A single intravitreal injection of 0.1 ml triamcinolone acetonide in a concentration of 4 mg / 0.1 ml.
  Interventions: Procedure: Intravitreal injection (4mg/0.1ml)
- Study group II: Suprachoroidal injection of full dose (Active Comparator): A single suprachoroidal injection of 0.1 ml triamcinolone acetonide in a concentration of 4 mg / 0.1 ml.
  Interventions: Procedure: Superachoroidal injection (4 mg/0.1ml)
- Study group III : Suprachoroidal injection of half dose (Active Comparator): They will receive a single suprachoroidal injection of 0.1 ml triamcinolone acetonide in a concentration of 2 mg / 0.1 ml.
  Interventions: Procedure: Suprachoroidal injection (2mg/0.1ml)

INTERVENTIONS:
Procedure: Intravitreal injection (4mg/0.1ml) — Injection will be performed in the operating room under complete sterile conditions Under topical anaesthesia. Intravitreal injection (4mg/0.1ml) of triamicinolone acetonide will be done using a 30-31 gauge needle at a distance of 3.5 mm from the limbus in aphakic or pseudophakic patients, and 4 mm in phakic patients. The needle will be then removed with application of cotton tipped applicator over the entry site.
  -IOP monitoring will be done at 15, 30 and 60 minutes following injection in all groups.
  Arms: Study group I : Intravitreal injection
Procedure: Superachoroidal injection (4 mg/0.1ml) — Injection will be performed in the operating room under complete sterile conditions Under topical anaesthesia. Suprachoroidal injection (4mg/0.1ml) of triamcinolone acetonide will be done using a custom-made 30-31 gauge needle with a sleeve to prevent further penetration of the needle into the vitreous cavity. Injection will be done at approximately 4 mm from the limbus.
  * IOP monitoring will be done at 15, 30 and 60 minutes following injection in all groups.
  * UBM assessment will be done 24 hours following injection to confirm targeting of the suprachoroidal space.
  Arms: Study group II: Suprachoroidal injection of full dose
Procedure: Suprachoroidal injection (2mg/0.1ml) — njection will be performed in the operating room under complete sterile conditions Under topical anaesthesia. Suprachoroidal injection (2mg/0.1ml) of triamcinolone acetonide will be done using a custom-made 30-31 gauge needle with a sleeve to prevent further penetration of the needle into the vitreous cavity. Injection will be done at approximately 4 mm from the limbus.
  * IOP monitoring will be done at 15, 30 and 60 minutes following injection in all groups.
  * UBM assessment will be done 24 hours following injection to confirm targeting of the suprachoroidal space.
  Arms: Study group III : Suprachoroidal injection of half dose

SUMMARY:
Intravitreal triamcinolone acetonide is a well-known method of treatment of diabetic macular edema, however, it has many side effects, most commonly causing cataract and glaucoma. Suprachoroidal route is an emerging route of delivery of intraocular drugs.

This is to our knowledge the first prospective study to compare the effect of triamcinolone acetonide delivered via the intravitreal versus the suprachoroidal route in the treatment of diabetic macular edema as regards safety and efficacy.

DETAILED DESCRIPTION:
The purposes of this study were:

1. To compare between intravitreal and suprachoroidalTA injection for treatment of DME in terms of improvement in both best corrected visual acuity (BCVA) and central macular thickness (CMT), and development of complications.
2. To identify which dose of TA will be efficient using the suprachoroidal route.

   * Type of Study: A prospective interventional randomized comparative study.
   * Study setting:Ophthalmology Department, Ain Shams University.
   * Study period:2 years.
   * Study population: Patients having DME.
   * Sample size: The study will be conducted on 45 eyes. This was done using PASS program, setting alpha error at 5% and power at 80%. Results from previous study (Koc et al., 2017) showed that the mean improvement in BCVA after 6 months of intravitreal injection of TA was 4.6 ± 8.8. While it is assumed to be 12.6 and 14.6 for the low dose and high dose suprachoroidal route.
   * Ethical considerations: Explanation of the procedure will be done for all patients and an informed written consent will be taken. Ethics committee approval will be obtained from the Institutional Review Board of the Faculty of Medicine, Ain Shams University.

All patients will undergo the following at initial presentation:

* Careful history taking.
* Full ophthalmological assessment including:

Baseline BCVA. Anterior segment examination using slit lamp biomicroscopy. IOP measurement using Goldmann applanation tonometer. Posterior segment examination using binocular indirect ophthalmoscopy and indirect slit lamp biomicroscopy (+90D Volk lens) for detailed evaluation of the macula and optic nerve head.

Fundus photography using VX-20 Kowa fundus camera, Japan. Ultrasound biomicroscopy (UBM) for measurement of scleral thickness in groups (II) and (III)using VuMax, Sonomed Escalon, theUnited States of America.

Spectral domain optical coherence tomography (SD-OCT) imaging using Retinascan RS 3000 advance, Nidek co.ltd, Gamgori, Japan.

Examination protocol: Macular map and 12 radial line scans to determine central macular thickness (1mm) and macular thickness in the inner 3 and 6 mm rings divided each into four quadrants.

Duration of follow up: 6 months.

Follow up schedule:

Follow up visits will be done at 1 day, 1 week, 1 month,3 months and 6 months.During the follow up, the following will be done:

* BCVA measurement.
* Full ophthalmological examination.
* Fundus photography after six months of injection.
* CMT measurement using SD-OCT at 1,3 and 6 months post-injection. In case of resistance to treatment (worsening of BCVA or CMT, or persistence of macular edema with central thickness less than 300µm), reinjection will be considered using the same drug and/or anti-VEGF agents.

ELIGIBILITY:
Inclusion Criteria:

* Type-II Diabetes Mellitus patients.
* Centrally involving DME with central thickness<300µm with no vitreomacular traction.
* Recently diagnosed DME or received treatment for DME in more than six months.

Exclusion Criteria:

* Pre-existingretinal disease other than diabetic retinopathy.
* Diabetic macular ischemia.
* IOP ≥ 21 mmHg and/or asymmetrical cup disc ratio or glaucoma patients.
* Prior cataract extraction of less than six months.
* Opaque media, uncooperative patients or patients with poor fixation.
* Any uncontrolled systemic disease.
* Systemic or local medicationsthat might affect the macular thickness

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-08-07 (Estimated); Study Completion 2021-08-07 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | Six months after injection
  Change in BCVA (Log.MAR) equal or more than 1 line

SECONDARY OUTCOMES:
Central macular thickness (CMT) | Six months after injection
  Change in CMT (um) equal or more than 50 um
Complications | During the six months after injection
  e.g. change in intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman G Salman, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt